CLINICAL TRIAL: NCT00656500
Title: Increasing QUITPLAN Helpline Utilization in Surgical Patients
Brief Title: Quitline Use in Surgical Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, David Warner, MD, Mayo Clinic
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 06-004330
Record Dates: First submitted 2008-04-04; First posted 2008-04-11 (Estimated); Last update posted 2012-02-03 (Estimated); Status verified 2012-02

CONDITIONS: Tobacco Dependence
Keywords: surgical patients; cigarette smoking; postoperative complications; telephone counseling; quitlines
MeSH Terms: conditions — Tobacco Use Disorder; Cigarette Smoking; Postoperative Complications

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Brief assistance with smoking abstinence
  Interventions: Behavioral: Standard brief advice
- 2 (Experimental): Brief intervention to promote quitline utilization
  Interventions: Behavioral: Quitline intervention

INTERVENTIONS:
Behavioral: Standard brief advice — Brief general assistance with smoking cessation
  Arms: 1
Behavioral: Quitline intervention — Brief intervention designed specifically to encourage quitline utilization
  Arms: 2

SUMMARY:
Elective surgery represents a teachable moment to deliver tobacco interventions. The overall goal of this proposal is to increase the utilization of the QUITPLANSM Helpline by surgical patients who smoke. Two specific aims will be pursued using a multidisciplinary research team. In the first aim, we will develop a practice-based intervention to promote QUITPLANSM Helpline utilization by surgical patients (Specific Aim 1A) using a combination of key informant interviews (approximately 30 subjects), and focus groups (approximately 25 subjects) then develop methods to educate providers in its implementation (Specific Aim 1B) and test their effectiveness in approximately 20 providers. In the second aim, we will perform a randomized clinical trial of this intervention in 300 patients scheduled for elective surgery, with the primary outcome being utilization of the QUITPLANSM Helpline (Specific Aim 2). Subjects will be randomized to receive either the intervention developed in Specific Aim 1, or a brief control intervention.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 18 yrs. scheduled for elective surgery at Mayo Clinic Rochester.
* Current smoking before the scheduling of surgery, defined as > 100 cigarettes lifetime consumption and self-reports of smoking either every day or some days. Patients who are in the midst of a quit attempt initiated since learning about surgery are eligible.

Exclusion Criteria:

* Patient is not available for telephone follow-up

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2007-07; Primary Completion 2010-02 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Completion of one quitline counseling session | Three months postoepratively

SECONDARY OUTCOMES:
Smoking behavior at six months postoperatively | six months postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: David O. Warner, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

REFERENCES:
- [Derived] Warner DO, Klesges RC, Dale LC, Offord KP, Schroeder DR, Shi Y, Vickers KS, Danielson DR. Clinician-delivered intervention to facilitate tobacco quitline use by surgical patients. Anesthesiology. 2011 Apr;114(4):847-55. doi: 10.1097/ALN.0b013e31820d868d. PMID 21317630